CLINICAL TRIAL: NCT06472986
Title: Feasibility and Efficacy of Activity-Based Therapy and Transcutaneous Spinal Cord Stimulation for Neurorestoration of Upper Limbs After Cervical Spinal Cord Injury
Brief Title: Activity-Based Therapy and Transcutaneous Spinal Cord Stimulation After Spinal Cord Injury (ABT-TCSCS)
Acronym: ABT-TCSCS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Ontario Neurotrauma Foundation (Other)
Responsible Party: Principal Investigator, Sukhvinder Kalsi-Ryan, Lead of the KITE Rehabilitation and Innovation Clinics-Lyndhurst Site, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-6276
Record Dates: First submitted 2024-06-18; First posted 2024-06-25 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Spinal Cord Injuries; Spinal Cord Injury Cervical
Keywords: stroke; cerebrovascular accident; CVA
MeSH Terms: conditions — Spinal Cord Injuries; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ABT-TCSCS (Experimental): The participants will receive activity-based therapy combined with transcutaneous spinal cord stimulation.
  Interventions: Other: Activity-based therapy and transcutaneous spinal cord stimulation

INTERVENTIONS:
Other: Activity-based therapy and transcutaneous spinal cord stimulation — Activity Based Therapy (ABT) is a method of neuro-rehabilitation that incorporates a high intensity, long duration and effortful engagement from the individual receiving therapy, to garner improvements in sensory and motor function. The ABT constitutes 4 types of exercises including: cardio-fitness, resistance, postural/weightbearing and functional exercises. TransCutaneous Spinal Cord Stimulation (TCSCS) stimulates spinal networks in the cervical region to neuro-modulate the descending motor commands/motor intentions from the brain, which control the muscles. In tCSCS, electrical stimulation is delivered at a frequency of 30-50Hz at 500-1000µs between C3-C7. 12 sessions of ABT (4 weeks), followed by 28 sessions of ABT-TCSCS (7 weeks). Each session will last 1 hour and delivered 3 times per week.

SUMMARY:
The ABT-TCSCS study investigates how feasible and beneficial are activity-based therapy and transcutaneous spinal cord stimulation on improving of arm and hand recovery after cervical spinal cord injury.

DETAILED DESCRIPTION:
The ABT-TCSCS is a one-arm interventional study evaluating the feasibility and efficacy of activity-based therapy and transcutaneous spinal cord stimulation on neurorestoration of upper limbs after cervical spinal cord injury. Up to 24 individuals with SCI who suffer from tetraplegia will be treated with ABT-TCSCS. All participants will receive 12 sessions of ABT (4 weeks), followed by 28 sessions of ABT-TCSCS (7 weeks). Each session will last 1 hour and delivered 3 times per week. All study participants will be assessed at the start of the study (Baseline 1) and then re-assessed after 6 weeks (Baseline 2) to ensure that they are neurologically stable. The baseline assessment will consist of the International Standards of Neurological Classification of SCI (ISNCSCI), GRASSP Version 1, the Spinal Cord Independence Measure (SCIM) and the TRI hand function test (TRI-HFT). Participants will be re-assessed after receiving 12 sessions of ABT i.e after 4 weeks (Pre-cervical stimulation assessment) and then after receiving 28 sessions of combined ABT and neuromodulation i.e after 7 weeks (Post-intervention assessment).

ELIGIBILITY:
Inclusion Criteria:

* Individuals with chronic traumatic and non-traumatic cervical SCI (ASIA classification A-incomplete**, B, C, D) between C1-C8
* Adults more than 18 years old
* At least 6 months post-spinal cord injury
* A score of 2 - 15 on the upper extremity motor score of the ISNCSCI
* A score between 5 - 40 on GRASSP Version 1 Strength on at least one side
* Individuals who are medically stable

Exclusion Criteria:

* Individuals with any other upper extremity deficit
* Unable to provide informed consent
* Unable to participate in an intensive rehabilitation outpatient program
* Spasticity that limits the range of motion greater than 50% for the elbow or wrist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-10-07 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
International Standards of Neurological Classification of SCI (ISNCSCI) | At enrollment, 4-6 weeks after enrollment, after 4 weeks (12 sessions) of ABT, and after 7 weeks (28 sessions) of ABT-TCSCS
  The ISNCSCI will be used to establish severity of injury, classify the sample and establish inclusion for study to be administered by clinicians. The ISNCSCI evaluates both motor and sensory impairment to determine the sensory and motor levels for the right and left side, the overall neurological level of the injury and completeness of the injury i.e. whether the injury is complete or incomplete. The severity of injury is graded as ASIA A = Complete, B (Sensory Incomplete), C (Motor Incomplete), D (Motor Incomplete), E (Normal).
Graded Redefined Assessment of Strength, Sensation and Prehension (GRASSP) Version 1 | At enrollment, 4-6 weeks after enrollment, after 4 weeks (12 sessions) of ABT, and after 7 weeks (28 sessions) of ABT-TCSCS
  The GRASSP Version 1 evaluates sensorimotor and prehension function of upper extremity impairment and hand function through three domains: Strength, Sensation and Prehension. It will be administered by clinicians and takes about 30-45 minutes to complete.
Spinal Cord Independence Measure (SCIM) | At enrollment, 4-6 weeks after enrollment, after 4 weeks (12 sessions) of ABT, and after 7 weeks (28 sessions) of ABT-TCSCS
  The SCIM is a measure of independence and defines how much gain in global function one makes.
TRI hand function test (TRI-HFT) | At enrollment, 4-6 weeks after enrollment, after 4 weeks (12 sessions) of ABT, and after 7 weeks (28 sessions) of ABT-TCSCS
  TRI-HFT will be used as a measure of functional and performance change before and after intervention.
Tactile Discrimination Test (TDT) | At enrollment, 4-6 weeks after enrollment, after 4 weeks (12 sessions) of ABT, and after 7 weeks (28 sessions) of ABT-TCSCS
  The TDT will be used to measure of ability to discriminate differences in finely graded texture.

SECONDARY OUTCOMES:
Neurophysiological Assessment using surface electromyography (EMG) | After 4 weeks (12 sessions) of ABT, and after 7 weeks (28 sessions) of ABT-TCSCS
  Neurophysiological Assessment using surface EMG will be used to determine the responses to ABT and TCSCS in multiple upper limb muscles. sEMG responses to cervical spinal stimulation will be recorded simultaneously in multiple upper limb muscles unilaterally on the 1) deltoid anterior, 2) deltoid posterior, 3) biceps brachii, 4) triceps brachii, 5) flexor carpi radialis, 6) extensor carpi radialis, 7) abductor pollicis brevis, and 8) first dorsal interosseous muscles.

CONTACTS AND LOCATIONS:
Overall Officials: Sukhvinder Kalsi-Ryan, Principal Investigator — Toronto Rehabilitation Institute
Locations (1):
- Toronto Rehabilitation Institute, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
We do not plan to share the data from this study with any researchers outside this study.

REFERENCES:
- [Result] Kirshblum S, Botticello A, Lammertse DP, Marino RJ, Chiodo AE, Jha A. The impact of sacral sensory sparing in motor complete spinal cord injury. Arch Phys Med Rehabil. 2011 Mar;92(3):376-83. doi: 10.1016/j.apmr.2010.07.242. PMID 21353822
- [Result] Marino RJ, Burns S, Graves DE, Leiby BE, Kirshblum S, Lammertse DP. Upper- and lower-extremity motor recovery after traumatic cervical spinal cord injury: an update from the national spinal cord injury database. Arch Phys Med Rehabil. 2011 Mar;92(3):369-75. doi: 10.1016/j.apmr.2010.09.027. PMID 21353821
- [Result] Kalsi-Ryan S, Curt A, Verrier MC, Fehlings MG. Development of the Graded Redefined Assessment of Strength, Sensibility and Prehension (GRASSP): reviewing measurement specific to the upper limb in tetraplegia. J Neurosurg Spine. 2012 Sep;17(1 Suppl):65-76. doi: 10.3171/2012.6.AOSPINE1258. PMID 22985372
- [Result] Kalsi-Ryan S, Riehm LE, Tetreault L, Martin AR, Teoderascu F, Massicotte E, Curt A, Verrier MC, Velstra IM, Fehlings MG. Characteristics of Upper Limb Impairment Related to Degenerative Cervical Myelopathy: Development of a Sensitive Hand Assessment (Graded Redefined Assessment of Strength, Sensibility, and Prehension Version Myelopathy). Neurosurgery. 2020 Mar 1;86(3):E292-E299. doi: 10.1093/neuros/nyz499. PMID 31792501
- [Result] Kapadia N, Zivanovic V, Verrier M, Popovic MR. Toronto rehabilitation institute-hand function test: assessment of gross motor function in individuals with spinal cord injury. Top Spinal Cord Inj Rehabil. 2012 Spring;18(2):167-86. doi: 10.1310/sci1802-167. PMID 23459270
- [Derived] Gopaul U, Bayley MT, Kalsi-Ryan S. Combined Activity-Based Therapy and Cervical Spinal Cord Stimulation: Active Ingredients, Targets and Mechanisms of Actions to Optimize Neurorestoration of Upper Limb Function After Cervical Spinal Cord Injury. Physiother Res Int. 2025 Apr;30(2):e70036. doi: 10.1002/pri.70036. PMID 39927575